CLINICAL TRIAL: NCT02274493
Title: Pilot Study of Robotic-Assisted Harvest of the Latissimus Dorsi Muscles
Brief Title: Robotic Harvest of the Latissimus Dorsi (LD) Muscles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0232; NCI-2015-00616 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Other Reconstructive Surgery; Failure of Muscle Graft; Cancer; Complications; Surgical Procedure, Unspecified
Keywords: da Vinci® robotic surgical system; latissimus dorsi muscle flap harvest procedures; breast reconstruction; scalp reconstruction; upper extremity reconstruction; lower extremity reconstruction
MeSH Terms: conditions — Neoplasms | interventions — Robotic Surgical Procedures; Plastic Surgery Procedures; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Robotic Harvest of the LD Muscles (Experimental): Surgical harvesting of the Latissimus Dorsi (LD) Muscles using da Vinci® robotic surgical system in participants undergoing LD muscle flap harvest procedures in conjunction with breast, scalp, upper extremity and lower extremity reconstructive surgery procedures.
  Interventions: Device: da Vinci® Robotic Surgical System; Procedure: LD muscle flap harvest procedure; Procedure: Reconstructive surgery; Behavioral: Questionnaires

INTERVENTIONS:
Device: da Vinci® Robotic Surgical System — Da Vinci Robotic Surgical system to be used in procedures that harvest the latissimus dorsi muscle for reconstructive procedures
  Other Names: Robotic surgery
Procedure: LD muscle flap harvest procedure — Latissimus dorsi muscle flap harvest procedure using da Vinci® Robotic Surgical System for use in reconstructive surgery.
Procedure: Reconstructive surgery — Reconstructive surgery is considered to be standard of care.
Behavioral: Questionnaires — Questionnaire about pain, as well as participant's shoulder, arm, and hand range of motion completed at baseline, and at follow up visits 3-6.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to learn more about the safety and feasibility of using the Da Vinci Robotic Surgical system in procedures that harvest the latissimus dorsi muscle (a back muscle below your shoulder) for reconstructive procedures.

DETAILED DESCRIPTION:
If participant is found to be eligible to take part in this study, and participant agrees, participant's screening, reconstructive surgery, and follow-up appointments will be scheduled over multiple visits, as listed in this consent form. All procedures will be performed on days in which standard of care procedures would already be performed.

If it is determined that participant is eligible, the following will be performed before the surgery:

* The study doctor or a member of the research team will review participant's medical information and ask participant questions about participant's medical history and demographic information.
* Participant will have a physical exam.
* Participant will be evaluated by a Physical Therapist to test participant's range of motion and strength.
* Participant will complete a questionnaire about pain, as well as participant's shoulder, arm, and hand range of motion. This information will be used to compare with the results after the surgery. This will take about 5 minutes to complete.
* Photographs and/or videos of the surgical site will be taken.
* If participant can become pregnant, participant will have a urine pregnancy test. To take part in this study, participant must not be pregnant.

Surgery Study Visit (2):

At this visit, participant's reconstructive surgery will be performed using a robot, called the Da Vinci® Robotic Surgical System. The reconstructive surgery is considered to be standard of care. Participant will be asked to sign a separate consent form that discusses the possible benefits and risks of the standard of care surgical procedure in more detail, including information about any anesthetic participant will be given for the surgery.

A standard muscle harvest procedure takes about 2 hours. A muscle harvest procedure with the robotic system is expected to take longer than the standard surgery. The total procedure time will vary for each patient depending on the type of muscle harvest procedure and other factors in the operating room. The total time to complete the muscle harvest and reconstruction will take about 4 hours. Photographs and/or videos of the surgical site will be taken.

Participant will remain in the hospital for 3-4 days after the surgery is complete for observation. After participant is discharged from the hospital, participant will need to return within 2 weeks for participant's first follow-up examination.

Follow-Up Study Visits (3-6):

After participant has been discharged from the hospital, participant will have 4 follow-up visits.

The first follow up visit will take place within two weeks after participant is discharged . The second follow-up visit will be between 2-4 weeks, the third follow up visit will be between 1-3 months and the fourth follow up will be between 3-6 months after participant is discharged.

The following tests and procedures will be performed at each follow-up visit:

* The study doctor will check the surgery site(s).
* Participant's overall health status will be checked.
* Participant will be evaluated by a Physical Therapist to test participant's range of motion and strength.
* Photographs and/or videos of the surgical site may be taken.
* Participant will complete the questionnaire about pain and participant's shoulder, arm, and hand range of motion. This information will be used to compare with the results from before the surgery.

Length of Study Participation:

Participation on the study will be over after the follow-up visits.

This is an investigational study. The use of the Da Vinci® Robotic Surgical System for surgery in the thorax (part of the upper body) is FDA approved and commercially available at this time. However, the system has not been FDA cleared specifically for use in latissimus dorsi muscle harvest procedures. The use of the DaVinci Robotic Surgical System for this type of reconstructive surgery has not been performed in live humans and is what researchers are investigating for this study.

Up to 15 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be equal to or greater than 18 years of age.
2. The subject must be willing and able to provide informed consent.
3. The subject is willing and able to comply with the study protocol.
4. The subject is undergoing one of the following reconstructive procedures that requires latissimus dorsi muscle harvest: a. Post-mastectomy breast reconstruction procedure (either nipple or skin sparing) in which a female subject needs additional muscle coverage over an implant, but does not need additional skin (i.e., patient is a candidate for a pedicled latissimus dorsi muscle flap procedure); b. Scalp reconstruction procedure in which the subject needs a free latissimus dorsi muscle flap for wound coverage; c. Upper extremity reconstruction procedure in which the subject needs a free latissimus dorsi muscle flap for wound coverage; or, d. Lower extremity reconstruction procedure in which the subject needs a free latissimus dorsi muscle flap for wound coverage.
5. The subject agrees to follow-up examinations out to 6 months post-treatment.

Exclusion Criteria:

1. The subject has a BMI > 35.
2. The subject has a history of significant bleeding disorders.
3. The subject is diabetic.
4. The subject is known or suspected to be pregnant or lactating.
5. The subject has a history of peripheral vascular disease.
6. The subject is a current smoker (has smoked within 4 weeks prior to surgery).
7. The subject has had prior back or axillary surgeries which could compromise the blood supply of the flap.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07-08 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C. Selber, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Latissimus Dorsi Muscle Harvest: Latissimus dorsi muscle harvest using the DaVinci robotic approach
Period: Overall Study
Arm/Group | Latissimus Dorsi Muscle Harvest
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Latissimus Dorsi Muscle Harvest
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 49.2 [28 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Latissimus dorsi muscle function [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Donor Site Complications and Muscle Flap Viability
Description: Muscle flap viability was determined by measuring the blood flow into and out of the muscle flap with a hand held Doppler after muscle harvest was complete
Time Frame: Participants were followed for up to a total of 6 months post-operatively
Population: All participants were assessed for the primary measure
Measure: Count of Participants; unit: Participants
Arm/Group | Latissimus Dorsi Muscle Harvest
Number analyzed (Participants) | 15
Participants | 15

2. Primary Outcome: Number of Participants With LD Muscle Flap Viability Following Robotic-Assisted Harvest Procedure
Time Frame: Participants were followed for up to a total of 6 months post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Latissimus Dorsi Muscle Harvest
Number analyzed (Participants) | 15
Participants | 15

3. Secondary Outcome: Evaluation of Donor Site Complications Through 6 Months Post-procedure
Description: The participants listed were evaluated for donor site complication.
Time Frame: Participants were followed for up to a total of 6 months post-operatively
Population: 1 participant withdrew study consent prior to post-procedure follow up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Latissimus Dorsi Muscle Harvest
Number analyzed (Participants) | 15
Participants | 14

4. Secondary Outcome: LD Muscle Flap Failure Through 6 Months Post-procedure
Description: Flap failure is defined as irreversible arterial and venous thrombosis detected by implantable or surface doppler signal.
Time Frame: Participants were followed for up to a total of 6 months post-operatively
Population: 1 participant withdrew study consent prior to post-procedure follow up visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Latissimus Dorsi Muscle Harvest
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: Subjects were followed for a total of 6 months post-operatively
Arm/Group | Latissimus Dorsi Muscle Harvest
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Latissimus Dorsi Muscle Harvest (N=15)
Infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Latissimus Dorsi Muscle Harvest (N=15)
Infection (Infections and infestations) | 1
Seroma (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT02274493/Prot_SAP_000.pdf